CLINICAL TRIAL: NCT03294733
Title: The Relationship Between Age and Carpal Tunnel Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter M. Murray, Chair, Orthopedic Department Mayo Clinic Florida, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-002345
Record Dates: First submitted 2017-09-19; First posted 2017-09-27 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Carpal Tunnel
MeSH Terms: conditions — Median Neuropathy | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: ultrasound carpal tunnel size on subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Other): Ultrasound wrists to determine carpal tunnel size
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — This ultrasound machine is owned by the department of orthopaedic surgery and is capable of up to 15 MHz image definition with its linear transducer

SUMMARY:
Investigators hypothesis is that as human age increases, the size of the carpal tunnel decreases.

DETAILED DESCRIPTION:
Participants will be taken to a hand examination room where a portable ultrasound (US) machine is present. A previously determined wrist will be examined for each of the participants. The US will be used to obtain measurements of the subjects carpal tunnel and median nerve at multiple levels in order to define its size.

ELIGIBILITY:
Inclusion Criteria:

* Greater than age 18 having bilateral wrists amenable to ultrasound examination.

Exclusion Criteria:

* Active carpal tunnel syndrome,
* history of carpal tunnel syndrome
* any prior arm or hand surgery (including previous carpal tunnel release for any reason or previous surgery on the volar wrist)
* distal radius fracture deformity
* rheumatoid arthritis
* open wounds or lesions of the hand or forearm
* known congenital deformities of the upper extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Size of carpal tunnel | Baseline
  using ultrasound imaging to determine size of carpal tunnel

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Murray, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials